CLINICAL TRIAL: NCT00799240
Title: MK-0646 IMPACT Study: MK-0646, Insulin Growth Factor 1 Receptor Antibody in Stage IIIB or IV Metastatic Non-Squamous Lung Cancer, Combined With Pemetrexed (Alimta) and Cisplatin, a Randomized Phase II Trial.
Brief Title: MK-0646 Insulin Growth Factor 1 Receptor Antibody in Stage IIIb or IV Metastatic Non-Squamous Lung Cancer
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11386; MK-0646 (Other: Merck)
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; stage IIIb; pleural effusion; stage IV; metastatic lung cancer; non squamous lung cancer; IGF-1R; Pemetrexed; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Pleural Effusion; Insulin-Like Growth Factor I, Resistance To | interventions — dalotuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A Pemetrexed Cisplatin (Active Comparator): Arm A: Pemetrexed, cisplatin: pemetrexed and cisplatin chemotherapy at standard doses given IV every 21 days. Patients will be treated for a maximum of 6 cycles.
  Interventions: Drug: Arm A: Pemetrexed Cisplatin
- Arm B Permetrexed, Cisplatin, MK-0646 (Experimental): Pemetrexed and cisplatin chemotherapy at standard doses given IV every 21 days in combination with MK-0646 given IV, 10 mg/Kg, Days 1, 8 and 15 weekly
  Interventions: Drug: Arm B Pemetrexed, Cisplatin and MK-0646

INTERVENTIONS:
Drug: Arm A: Pemetrexed Cisplatin — Pemetrexed: 500mg/m2 IV on day 1 and Cisplatin: 75 mg/m2 IV on day 1 every 21 days x 6 cycles.
  Other Names: MK-0646
  Arms: Arm A Pemetrexed Cisplatin
Drug: Arm B Pemetrexed, Cisplatin and MK-0646 — Pemetrexed 500 mg/m2 IV on Day 1 and Cisplatin 75 mg/m2 IV on Day 1 every 21 days for 6 cycles in combination with MK-0646 will be given IV, 10 mg/KG, Days 1, 8 and 15 weekly.
  Other Names: MK-0646
  Arms: Arm B Permetrexed, Cisplatin, MK-0646

SUMMARY:
This study will compare the rate of chemotherapy: pemetrexed and cisplatin compared with the combination of pemetrexed/cisplatin with MK-0646. The other purposes are to determine how long we can control the cancer growth and toxicity and safety of the combination. Laboratory research with the tumor tissue and blood obtained will be done to assess IGF-1R expression and related markers and correlate with response and survival.

DETAILED DESCRIPTION:
Insulin-like Growth factor 1 receptor (IGF-1R) is a tyrosine kinase receptor that regulates cell growth, proliferation and apoptosis.(4) Increased IGF1 signaling results in upregulation of proliferation and inhibition of apoptosis through RAF and PI3K pathways.(5) Several types of cancer, including non-small cell lung cancer, express IGF-1R and its ligand. The sequestration of IGF by IGF binding protein was associated with improved survival in patients with resected stage I lung cancer.(6) High expression of IGF-1R is associated with poor survival in surgically resected stage I lung cancer, specifically adenocarcinoma subtype. Patients with adenocarcinoma and never smoker had higher expression of IGF-1R vs. squamous cell carcinoma and smokers.(7). Low IGF-1R expression was associated with significant improvement in survival in the adenocarcinoma lung cancer but there was a lack of correlation between expression of IGF1R and survival in patients with squamous cell histology.

Monoclonal antibodies target the extracellular domain of IGF-IR and small molecules inhibit IGF-1R kinase. This is a potential new strategy in the treatment of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven newly diagnosed Stage IlIB or Stage IV advanced primary non-small cell bronchogenic lung cancer (non-squamous cell to include bronchoalveolar, adenocarcinoma, large cell carcinoma, or unspecified).
* clinically significant pleural effusion must have a thoracentesis.
* Patients with brain metastases are eligible provided they have completed brain radiation, neurologically stable, off dexamethasone for at least 1 week prior to registration. Patients with asymptomatic brain metastatic disease are eligible if they do not require radiation and are neurologically stable without dexamethasone.
* measurable disease documented by CT, MRI, X-ray or physical exam. Measurable disease must be assessed within 28 days prior to registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 28 days prior to registration. All disease must be assessed and documented.
* Prior radiation is permitted; at least one week must have elapsed since the completion of prior radiation therapy and must have recovered from all associated toxicities at time of registration. Measurable or non-measurable disease must be outside the previous radiation field or a new lesion must be present.
* At least 4 weeks have elapsed since surgery (thoracic or other major surgeries) and patients have recovered from all associated toxicities at the time of registration. Measurable disease must be present outside the area of surgical resection. There must be no anticipation of need for major surgical procedures during protocol treatment.
* Age ≥ 18 years old.
* ECOG performance status of 0-1.
* adequate bone marrow function defined by platelet count at least 100,000/mm3, hemoglobin ≥ 9g/dl, leukocyte count at least 3,000/mm OR absolute neutrophil count at least 1,500/mm3.
* adequate hepatic function documented by serum bilirubin ≤ 1.5x upper normal limit, AST or ALT, and alkaline phosphatase all ≤ 3 x IULN within 28 days prior to registration. (Except in presence of known hepatic metastasis, wherein AST or ALT may be up to 5 X upper normal limit.)
* serum creatinine ≤ institutional upper limit of normal (IULN) AND calculated or measured creatinine clearance ≥ 50 ml/mm using the Cockcroft Gault Formula. These tests must have been performed within 28 days prior to registration.
* ability to give informed consent.
* Able to provide consent for gene expression profiling, histopathology, and/or immunohistochemical assays
* Women of childbearing potential must have negative serum pregnancy test.
* Patients taking NSAIDs must agree to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed.
* ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.

Exclusion Criteria:

* Prior systemic chemotherapy or biologic therapy for non-small cell lung cancer. If neoadjuvant therapy or adjuvant therapy was given, patient must be at least 1 year out from the last chemotherapy and fully recovered from all toxicities.
* Cardiovascular: uncontrolled congestive heart failure, high blood pressure, unstable angina, or myocardial infarction within the prior year,serious cardiac arrhythmias requiring medication.
* Serious uncontrolled active infection, acute hepatitis or known HIV.
* Prior history of severe allergy (grade 3 or 4) to human monoclonal antibody.
* Concurrent use of human growth hormone or growth hormone inhibitors.
* Uncontrolled diabetes mellitus defined as a Hemoglobin A1C≥ 7.
* An other active malignancy in the past 2 years.
* Pregnant or nursing women are not eligible to participate in this trial due to the potential teratogenic or abortifacient effects of the study drug on the fetus or nursing infant. Persons of reproductive potential must have agreed to use two methods of effective contraception prior to, during, and for 4 weeks after study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Compare response rate between the two arms. | 31 months

SECONDARY OUTCOMES:
Progression-free survival, overall survival and Toxicity profile | 31 months
Exploratory Objectives: Assess biomarkers of Pemetrexed, IGF-1R and immunogenicity of MK-0646. | 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Chao H Huang, MD, FACP, Principal Investigator — University of Kansas Medical Center
Locations (4):
- United States (4):
  - Hutchinson Clinic, PA, Hutchinson, Kansas
  - Kansas University Cancer Center, Kansas City, Kansas
  - Stormont Vail Healthcare, Topeka, Kansas
  - VA Medical Center, Kansas City, Missouri

REFERENCES:
- [Derived] Huang CH, Williamson SK, Neupane P, Taylor SA, Allen A, Smart NJ, Uypeckcuat AM, Spencer S, Wick J, Smith H, Van Veldhuizen PJ, Kelly K. Impact Study: MK-0646 (Dalotuzumab), Insulin Growth Factor 1 Receptor Antibody Combined with Pemetrexed and Cisplatin in Stage IV Metastatic Non-squamous Lung Cancer. Front Oncol. 2016 Jan 13;5:301. doi: 10.3389/fonc.2015.00301. eCollection 2015. PMID 26793618